CLINICAL TRIAL: NCT05516121
Title: An Open Non-comparative Clinical Trial of the Pharmacokinetics, Safety and Tolerability of VLT-015, Tablets, 100 mg (Valentech LLC) With Single and Multiple Use in Patients With Schizophrenia
Brief Title: VLT-015 in Patients With Schizophrenia
Acronym: VLT-015
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CF Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KI-VLT-001
Record Dates: First submitted 2022-07-22; First posted 2022-08-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: pharmacokinetic parameters; tolerability; safety; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): Each patient takes 100 mg single dose, after wash-out period 200 mg single dose, then, after wash-out period 200 mg single dose two following days
  Interventions: Drug: VLT-015

INTERVENTIONS:
Drug: VLT-015 — 100 mg single dose, 200 mg single dose, 200 mg single dose once a day for two consecutive days
  Other Names: FAP-2015

SUMMARY:
15 stable patients diagnosed with schizophrenia take 100 mg of VLT-015 once a day, 200 mg of VLT-015 once a day and 200 mg of VLT-015 on two consecutive days with an interval of 24 hours between doses. PK parameters are measured, tolerability and safety of the product are evaluated.

DETAILED DESCRIPTION:
At stage 1, 15 stable patients diagnosed with schizophrenia take 1 tablet of VLT-015 (100 mg) followed by blood sampling to measure the level of the active substance and its main metabolite within 72 hours. After that patients have 3 days washout period.

At the second stage, the same 15 patients take two 100 mg tablets of VLT-015 (200 mg) followed by blood sampling to measure the level of the active substance and its main metabolite within 72 hours. Then patients have the same 3 days washout period.

At stage 3, the same patients take 2 tablets of VLT-015 (200 mg) consecutively for 2 days with 24-hours interval followed by blood sampling to measure the level of the active substance and its main metabolite within 96 hours.

PK parameters are measured, tolerability and safety of the product are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 to 50
* Availability of a voluntarily signed Information Consent (Patient Information Sheet) for participation in this clinical research and further hospitalization;
* The diagnosis of schizophrenia established in the anamnesis
* The patient's stay in remission** based on the decision of the investigator before and after the withdrawal of maintenance therapy.

Criteria determining the state of remission:

* the sum of points of the Positive and Negative Symptom Scale (PANSS) according to positive Marder factor is less than 22 points,
* each item score of the positive Marder factor (delusions, hallucinatory behavior, grandiosity, suspicion, stereotyped thinking, somatic anxiety, unusual thought content, decreased criticism) less than 4 points

  * Absence of taking antipsychotic drugs for 5 periods half-life of the drug taken;
  * The patient's ability to adequately cooperate (the ability to understand provided information about the clinical trial, readiness for compliance with the requirements of the study protocol);
  * Agree to use barrier methods of contraception during the study and within 2 months after completion of the study.

Exclusion Criteria:

1. The presence of contraindications to the use of VLT-015:

   * dysfunction of the bone marrow;
   * hypersensitivity to VLT-015 and other components of the drug;
   * toxic or idiosyncratic granulocytopenia/agranulocytosis in history;
   * epilepsy;
   * alcohol, drug intoxication and coma;
   * collapse, depression of the central nervous system of any etiology;
   * severe kidney or heart disease;
   * paralytic intestinal obstruction;
   * glucose-galactose malabsorption;
   * renal or hepatic insufficiency;
2. Patients requiring medication or other concomitant therapies listed in the unacceptable concomitant therapy section;
3. The presence of prostatic hyperplasia or glaucoma in patients;
4. Diseases of the bone marrow in history;
5. Active tuberculosis, cystic fibrosis, systemic connective tissue diseases, oncological processes of any localization;
6. Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen the prognosis patient, and also make it impossible to conduct a clinical trial);
7. Alcoholism and drug addiction at the present time, or in history;
8. Lack of patient willingness to cooperate, non-compliance of the patient;
9. Participation of the patient in any other clinical study in the last 30 days;
10. Patients planning to stay in the hospital during the study period for reasons other than the purposes of this clinical trial.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Cmax | 3 weeks
  Maximum plasma concentration
Tmax | 3 weeks
  Time to reach the maximum concentration
AUC o-t | 3 weeks
  Area under the pharmacokinetic curve, starting from time zero until the time of last blood sample collection
AUC o - ∞ | 3 weeks
  Area under the pharmacokinetic curve, starting from time zero to infinity
AUC o-t/AUC o-∞ | 3 weeks
  Share of AUC o-t of AUC o-∞ expressed in %
T1/2 | 3 weeks
  Half-life, determined by the formula T_(1/2)= (ln⁡(2))/K_el
MRT | 3 weeks
  Mean retention time of the drug in the body, calculated from the start of the first time point to the time the last blood sample was taken

CONTACTS AND LOCATIONS:
Overall Officials: Max E Zapolski, Study Director — Valentech LLC
Locations (2):
- Russia (2):
  - Federal State Budgetary Scientific Institution "Mental Health Research Centre", Moscow, Moscow Oblast
  - GBUZ SK Stavropol Regional Clinical Specialized Psychiatric Hospital No. 1, Stavropol, Stavropol Oblast

IPD SHARING:
Plan to Share IPD: No